CLINICAL TRIAL: NCT03618134
Title: Phase Ib/II Trial of Stereotactic Body Radiotherapy (SBRT) in Cominbation With Immunotherapy Prior to Transoral Robotic Surgery (TORS) for Human Papillomavirus Positive (HPV+) Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Stereotactic Body Radiation Therapy and Durvalumab With or Without Tremelimumab Before Surgery in Treating Participants With Human Papillomavirus Positive Oropharyngeal Squamous Cell Caner
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001204; NCI-2018-01214 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-07-12; First posted 2018-08-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC (American Joint Committee on Cancer) v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Human Papillomavirus Positive; Oropharyngeal Squamous Cell Carcinoma; p16 Positive Neoplastic Cells Present; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Immunoglobulin G; Disulfides; Radiosurgery; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort I (SBRT, durvalumab, TORS, neck dissection) (Experimental): Beginning day 0 of course 1, participants undergo stereotactic body radiation therapy 5 days a week for 1 week and receive durvalumab IV over 1 hour on days 0 and 27 in the absence of disease progression or unacceptable toxicity. Participants then undergo transoral robotic surgery and modified radical neck dissection between weeks 6-8. Beginning week 12, participants then receive durvalumab IV over 1 hour every 4 weeks. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Procedure: Modified Radical Neck Dissection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy; Procedure: Transoral Robotic Surgery
- Cohort II (SBRT, durvalumab,tremelimumab,TORS,neck dissection) (Experimental): Beginning day 0 of course 1, participants undergo stereotactic body radiation therapy 5 days a week for 1 week and receive tremelimumab IV and durvalumab IV over 1 hour on days 0 and 27 in the absence of disease progression or unacceptable toxicity. Participants then undergo transoral robotic surgery and modified radical neck dissection between weeks 6-8. Beginning week 12, participants then receive durvalumab IV over 1 hour every 4 weeks. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Procedure: Modified Radical Neck Dissection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy; Procedure: Transoral Robotic Surgery; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Procedure: Modified Radical Neck Dissection — Undergo modified radical neck dissection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Procedure: Transoral Robotic Surgery — Undergo TORS
  Other Names: TORS
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
  Arms: Cohort II (SBRT, durvalumab,tremelimumab,TORS,neck dissection)

SUMMARY:
This phase Ib/II trial studies the side effects and how well stereotactic body radiation therapy and durvalumab with or without tremelimumab before surgery work in treating participants with human papillomavirus positive oropharyngeal squamous cell cancer. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Monoclonal antibodies, such as durvalumab and tremelimumab, may interfere with the ability of tumor cells to grow and spread. Giving stereotactic body radiation therapy and durvalumab with or without tremelimumab before surgery may work better in treating participants with oropharyngeal squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability associated with the following treatment regimens: Cohort 1: stereotactic body radiation therapy (SBRT) and durvalumab, followed by transoral robotic surgery (TORS) and adjuvant durvalumab and cohort 2: SBRT and durvalumab + tremelimumab, followed by TORS and adjuvant durvalumab. (Phase I safety lead-in) II. To assess the efficacy of the treatment combination deemed safe from Phase I in terms of progression free survival, in order to determine the non-inferiority of tumor control (progression-free survival [PFS] of 85% at 2 years) compared to conventional large field adjuvant radiotherapy +/- concurrent chemotherapy. (Phase II) III. To determine Common Terminology Criteria for Adverse Events (CTCAE) grade 3+ acute and chronic toxicities at the end of radiation, after surgery, at the end of adjuvant immunotherapy infusion, at 3 month, at 6 month, at 1 year, and at 2 years. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the objective response rate to durvalumab +/- tremelimumab + SBRT prior to TORS.

II. To determine the rate of subclinical lymph node involvement at time of TORS and neck dissection.

III. To determine the rate of contra-lateral neck failure with medial oropharyngeal and base of tongue primary lesions.

IV. To determine the potential salvage rate. V. To determine the locoregional control, distant control, and overall survival.

VI. To determine the incidence of all toxicity associated with treatment protocol.

VII. To determine the short- and long-term quality of life of patients on protocol.

TRANSLATIONAL OBJECTIVES:

I. To evaluate the impact of KRAS gene-variant mutation on immune response and treatment outcome.

II. To evaluate the impact of PI3K gene mutation on immune response and treatment outcome.

III. Saliva samples to evaluate biomarkers for immune response to human papillomavirus (HPV) associated oropharyngeal squamous cell carcinoma (OPSCC) to be collected prior to treatment, at time of TORS, and at each yearly follow-up visit.

IV. Blood samples to evaluate biomarkers of immune response to HPV associated OPSCC to be collected prior to treatment, at time of TORS, and at each yearly follow-up visit.

V. Tumor tissue taken at the time of initial biopsy and at time of resection will be profiled for tumor infiltrating lymphocytes; activation markers and antigen specific T-cell receptor (TCR) utilization/diversity will be evaluated for additional checkpoint targets.

VI. On long-term follow-up, tumor antigen specific T lymphocyte memory populations will be monitored for representation and robustness in in-vitro stimulation assays as potential biomarker of continued anti-tumor activity.

VII. Immortalization of tumor infiltrating B-cells for identification of antigen presenting complex, antibody specificity, and potential serologic markers of continuing long-term immune response in patients.

OUTLINE: Participants are assigned to 1 or 2 cohorts.

COHORT I: Beginning day 0 of course 1, participants undergo stereotactic body radiation therapy 5 days a week for 1 week and receive durvalumab intravenously (IV) over 1 hour on days 0 and 27 in the absence of disease progression or unacceptable toxicity. Participants then undergo transoral robotic surgery and modified radical neck dissection between weeks 6-8. Beginning week 12, participants then receive durvalumab IV over 1 hour every 4 weeks. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

COHORT II: Beginning day 0 of course 1, participants undergo stereotactic body radiation therapy 5 days a week for 1 week and receive tremelimumab IV and durvalumab IV over 1 hour on days 0 and 27 in the absence of disease progression or unacceptable toxicity. Participants then undergo transoral robotic surgery and modified radical neck dissection between weeks 6-8. Beginning week 12, participants then receive durvalumab IV over 1 hour every 4 weeks. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 12 weeks for 2 years and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluation.
* Pathologically proven diagnosis of HPV-positive squamous cell carcinoma of the oropharynx. HPV-positivity will be defined as tumors that are p16-positive by immunohistochemistry.
* Patients must have T0-3 disease with all gross disease amenable to R0 resection (reviewed by multidisciplinary study team) and is eligible for TORS in the opinion of the treating physician.
* N0-N2b with all cervical disease confined to 2 cervical lymph node levels if the involved nodal levels are adjacent.
* Karnofsky performance status >= 70.
* Body weight >= 50 kg.
* Patients who are medically operable, without pre-existing medical conditions that could inhibit surgery following neoadjuvant therapy, and do not refuse surgery.
* Patients with smoking history (< 20 pack year history) is allowed.
* Patients must have MRI neck with and without contrast and a diagnostic positron emission tomography (PET), computed tomography (CT) or PET/CT skull base to mid-thigh with contrast within 30 days prior to SBRT.
* Hemoglobin >= 9.0 g/dL.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3).
* Platelet count >= 100 (or 75) x 10^9/L (>= 75,000 per mm^3).
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert?s syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal.
* Serum creatinine > 40 mL/min.
* Female patients with reproductive potential (e.g., females menopausal for less than 1 year and not surgically sterilized) must agree to practice two highly effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of durvalumab monotherapy or for at least 180 days after completion of durvalumab/tremelimumab combination therapy. Female patients of childbearing potential must provide a negative pregnancy test (urine) prior to treatment initiation. Male patients, whose partners are women with reproductive potential, and the women themselves also must agree to practice two effective contraceptive measures.
* Female patients with evidence of post-menopausal status if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Karnofsky performance status (KPS) < 70.
* Body weight < 50 kg.
* Histology other than squamous cell carcinoma.
* Primary site other than oropharynx (i.e. oral cavity, salivary glands, nasal cavity, paranasal sinuses, larynx, or nasopharynx) or of unknown primary.
* Patients with synchronous or bilateral disease.
* Patient with N3 nodal disease, N2c nodal disease, and N2b disease with gross disease in more than 2 neck levels (levels not adjacent to each others are also not allowed).
* Patients with recurrent head and neck cancer.
* Patients with metastatic disease on initial staging study.
* Patients who underwent attempted resection rather than the diagnostic biopsy of the primary site or nodal sampling of the neck disease.
* Prior systemic therapy (chemotherapy, biologic, or immunotherapy) for the same OPSCC.
* Previous treatment with Anti-CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) including tremelimumab or PD1/PD-L1 inhibitor (programmed cell death) , including durvalumab.
* Concurrent enrollment in another clinical trial.
* Patients that received prior radiotherapy that would result in overlap of radiation therapy fields.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no evidence of active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease.
* Any concurrent anticancer therapy.
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from a baseline electrocardiogram using Fredericia?s correction.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone.
* History of allogeneic organ transplant.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, seizures, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, active peptic ulcer disease or gastritis, serious chronic gastrointestinal (GI) conditions associated with diarrhea, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ two highly effective birth control methods from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of investigational product (IP). Note: Local surgery of isolated lesions for palliative intent is acceptable.
* Any unresolved toxicity National Cancer Institute (NCI) CTCAE grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study physician.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Known allergy or hypersensitivity to IP or any excipient.
* Subjects with uncontrolled seizures.
* History of leptomeningeal carcinomatosis.
* History of active primary immunodeficiency.
* Clinical documentation of active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase I safety lead-in) assessed Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.03 criteria | Up to 90 days after last dose
  Data from all cycles of treatment will be combined in the presentation of safety data. AEs will be listed individually by patient.
Progression-free survival (PFS) (Phase II) | From time of enrollment to the first occurrence of disease progression as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 or death from any cause, assessed up to 2 years
  The Kaplan-Meier product-limit estimate of the PFS function will be estimated and displayed. The median PFS time will be given with 95% confidence interval. Summaries of the number and percentage of patients experiencing a PFS event, and the type of event (RECIST v 1.1 or death) will be provided.
Incidence of grade >= adverse events (Phase II) | Up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of enrollment to date of death due to any cause, assessed up to 2 years
  OS will be estimated by Kaplan-Meier estimate. Summaries of the number and percentage of patients who have died, are still in survival follow-up, are lost to follow-up and have withdrawn consent will be provided along with median OS.
Primary tumor control determined by RECIST v. 1.1 | Up to 2 years
  Kaplan-Meier estimate will be used to describe primary tumor control rate.
Distant recurrence rate | Up to 2 years
  Distant recurrence rate will be determined by surveillance imaging, with failure defined as the appearance of new distant disease from the date of enrollment. Kaplan-Meier estimate will be used to describe distant recurrence rate.
Locoregional control rate | Up to 2 years
  Locoregional control rate will be determined by surveillance imaging, with failure defined as the appearance of new locoregional disease from the date of enrollment. Kaplan-Meier estimate will be used to describe locoregional control rate.
Rate of contralateral neck failure | Up to 2 years
  Will be determined by surveillance imaging, with failure defined as the appearance of new cervical lymphadenopathy from the date of enrollment. Kaplan-Meier estimate will be used to describe rate of contralateral neck failure.
Rate of subclinical lymph node involvement | At time of surgery
  Will be determined by surgical pathology findings.
Objective response rate | Up to 2 years
  The objective response rate will be determined by pre-surgical magnetic resonance imaging.
Incidence of adverse events assessed by CTCAE v4 | Up to 2 years
  The safety analysis set will be used for safety analyses. The overall safety and tolerability will be assessed throughout the study period. All adverse event data will be listed individually by treatment group and patient identifier.
Short quality of life | Up to 2 years
  Will be using the University Washington's Quality of Life Questionnaire (UW-QOL) v4. Assessment at baseline, with each cycle, post-stereotactic body radiation therapy, post-surgically, and throughout adjuvant therapy on a standard schedule. The scale is 0 (worst) to 100 (best)
long-term quality of life | Up to 2 years
  Will be using the Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN) version 4. questionnaire. Assessment at baseline, with each cycle, post-stereotactic body radiation therapy, post-surgically, and throughout adjuvant therapy on a standard schedule. The scale is 0 to 40. The higher the score the better quality of life (QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States